CLINICAL TRIAL: NCT04223752
Title: A Phase 1, Open-label, Non-comparative, Multicenter Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Ceftolozane/Tazobactam (MK-7625A) in Pediatric Participants With Nosocomial Pneumonia
Brief Title: Safety and Pharmacokinetics of Ceftolozane/Tazobactam in Pediatric Participants With Nosocomial Pneumonia (MK-7625A-036)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-036; MK-7625A-036 (Other: MSD Protocol Number); 2022-501110-56-00 (Registry Identifier: EU CT); U1111-1279-4959 (Registry Identifier: UTN); 2018-004704-19 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Nosocomial Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age (Experimental): Participants 12 to <18 years of age with nosocomial pneumonia receive intravenous (IV) ceftolozane/tazobactam every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/Tazobactam
- Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age (Experimental): Participants 7 to <12 years of age with nosocomial pneumonia receive IV ceftolozane/tazobactam every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/Tazobactam
- Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age (Experimental): Participants 2 to <7 years of age with nosocomial pneumonia receive IV ceftolozane/tazobactam every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/Tazobactam
- Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age (Experimental): Participants 3 months to <2 years of age with nosocomial pneumonia receive IV ceftolozane/tazobactam every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/Tazobactam
- Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age (Experimental): Participants from birth to <3 months of age with nosocomial pneumonia receive IV ceftolozane/tazobactam every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/Tazobactam

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam — Participants 12 to <18 years of age: IV ceftolozane 2 g with tazobactam 1 g infused over a 60-minute period.
  Participants <12 years of age: IV ceftolozane 40 mg/kg with tazobactam 20 mg/kg infused over a 60-minute period (not to exceed a dose of ceftolozane 2g and tazobactam 1 g).
  Other Names: MK-7625A

SUMMARY:
This is a phase 1, open-label, non-comparative, multicenter clinical study to evaluate the safety, tolerability, and pharmacokinetics of ceftolozane/tazobactam (MK-7625A) in pediatric participants with nosocomial pneumonia (NP).

ELIGIBILITY:
Inclusion Criteria:

* Is hospitalized and anticipated to receive a minimum of 8 days of concomitant standard-of-care [SOC] antibiotic therapy for proven or suspected NP.
* If male, is abstinent from heterosexual intercourse, or agrees to use contraception during the intervention period and for ≥30 days after the last dose of study intervention.
* If female, is not pregnant or breastfeeding, or is not a woman of childbearing potential (WOCBP), or is a WOCBP using acceptable contraception, is a WOCBP with negative urine or serum pregnancy test within 48 hours of the first dose of study intervention, or is abstinent from heterosexual intercourse.

Exclusion Criteria:

* Has a documented history of any moderate or severe hypersensitivity (or allergic) reaction to any β-lactam antibacterial.
* Participants 3 months to <18 years of age: has moderate to severe impairment of renal function, defined as an estimated creatinine clearance (CrCL) <50 mL/min/1.73 m2 based on the revised Schwartz equation or requirement for peritoneal dialysis, hemodialysis, or hemofiltration.
* Participants <3 months of age: has CrCL <20 mL/min/1.73 m2 based on the revised Schwartz equation or requirement for peritoneal dialysis, hemodialysis, or hemofiltration.
* Is receiving or is anticipated to receive piperacillin/tazobactam while receiving ceftolozane/tazobactam or has received piperacillin/tazobactam within 24 hours prior to the first dose of ceftolozane/tazobactam.
* Has participated in any clinical study of a therapeutic investigational product within 30 days prior to the first dose of ceftolozane/tazobactam.
* Has previous participation in any study of ceftolozane or ceftolozane/tazobactam.
* Has any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of study data.
* Has any rapidly progressing disease or immediately life-threatening illness including acute hepatic failure or septic shock.
* Has active immunosuppression.

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- United States (6):
  - AdventHealth Orlando ( Site 1318), Orlando, Florida
  - Mayo Clinic in Rochester, Minnesota ( Site 1322), Rochester, Minnesota
  - Montefiore Medical Center [Bronx, NY] ( Site 1313), New York, New York
  - Sanford Children's Hospital ( Site 1301), Sioux Falls, South Dakota
  - West Virginia University ( Site 1310), Morgantown, West Virginia
  - Children's Wisconsin ( Site 1321), Milwaukee, Wisconsin
- Hospital Roberto del Río ( Site 1400), Santiago, Region M. de Santiago, Chile
- Colombia (4):
  - Hospital General de Medellin ( Site 1503), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 1501), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 1500), Barranquilla, Atlántico
  - Oncomédica S.A.S ( Site 1506), Montería, Departamento de Córdoba
- Estonia (2):
  - SA Tallinna Lastehaigla/Tallinn Children's Hospital ( Site 0201), Tallinn, Harju
  - SA Tartu Ulikooli Kliinikum Lastekliinik ( Site 0200), Tartu, Tartu
- Hippokration General Hospital of Thessaloniki ( Site 0400), Thessaloniki, Central Macedonia, Greece
- Mexico (2):
  - Instituto Nacional de Pediatria-Unidad de Apoyo a la Investigación Clínica ( Site 1602), Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez-Infectious Diseases ( Site 1600), Mexico City, Mexico City
- Russia (3):
  - Morozovskaya Children City Clinical Hospital ( Site 0901), Moscow, Moscow
  - St. Olga Children City Hospital ( Site 0906), Saint Petersburg, Sankt-Peterburg
  - Smolensk Regional Clinical Hospital ( Site 0903), Smolensk, Smolensk Oblast
- Hospital Universitario Sant Joan de Deu ( Site 1100), Esplugues de Llobregat, Barcelona, Spain
- Ukraine (4):
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 1205), Dnipro, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Children Clinical Hospital ( Site 1204), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kharkiv City Children Hospital 16 ( Site 1200), Kharkiv, Kharkivs’ka Oblast’
  - Institution of Pediatr Obstetr and Gynec NAMS of Ukraine ( Site 1203), Kyiv, Kyivska Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26192&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled in error in the Group 5 arm and was excluded from the All participants as treated (APaT) population; the participant did not receive study intervention.
Groups:
- Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age: Participants 12 to <18 years of age with nosocomial pneumonia received intravenous (IV) ceftolozane 2g and tazobactam 1g every 8 hours for 8-14 days.
- Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age: Participants 7 to <12 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age: Participants 2 to <7 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age: Participants 3 months to <2 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age: Participants from birth to <3 months of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and 20 mg/kg tazobactam every 8 hours for 8-14 days.
Period: Overall Study
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Started | 8 | 7 | 8 | 10 | 8
Treated | 8 | 7 | 8 | 10 | 7
Completed | 8 | 7 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 2 | 2
Not completed — Participant enrolled in error | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age | Total
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 8 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.345 (1.6408) | 9.709 (1.9100) | 3.185 (0.7430) | 0.806 (0.2994) | 0.102 (0.0628) | 5.294 (5.6787)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 6 | 2 | 3 | 19
  Male | 2 | 5 | 2 | 8 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 3 | 3 | 3 | 15
  Not Hispanic or Latino | 7 | 2 | 5 | 7 | 5 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 7 | 4 | 7 | 7 | 5 | 30
  More than one race | 1 | 2 | 1 | 0 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants experiencing any AE was reported for each arm.
Time Frame: Up to 31 days
Population: The analysis population consisted of participants who received any dose (including partial doses) of ceftolozane/tazobactam.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 7
Percentage of participants | 50.0 (15.7) [15.7 to 84.3] | 71.4 (29.0) [29.0 to 96.3] | 75.0 (34.9) [34.9 to 96.8] | 90.0 (55.5) [55.5 to 99.7] | 85.7 (42.1) [42.1 to 99.6]

2. Primary Outcome: Percentage of Participants With Any Serious AEs (SAEs)
Description: An SAE was defined as any untoward medical consequence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other important medical event. The percentage of participants with any SAE was reported for each arm.
Time Frame: Up to 31 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 7
Percentage of participants | 12.5 (0.3) [0.3 to 52.7] | 28.6 (3.7) [3.7 to 71.0] | 0.0 (0.0) [0.0 to 36.9] | 30.0 (6.7) [6.7 to 65.2] | 28.6 (3.7) [3.7 to 71.0]

3. Primary Outcome: Percentage of Participants With Any Drug-related AEs
Description: A drug-related AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, and considered related to the study intervention. The percentage of participants with any drug related AEs was reported for each arm.
Time Frame: Up to 31 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 7
Percentage of participants | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 41.0] | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 30.8] | 14.3 (0.4) [0.4 to 57.9]

4. Primary Outcome: Percentage of Participants With Any Drug-related SAEs
Description: A drug-related SAE was defined any untoward medical consequence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other important medical event, that is considered related to the study intervention. The percentage of participants with any drug related SAEs was reported for each arm.
Time Frame: Up to 31 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 7
Percentage of participants | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 41.0] | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 30.8] | 0.0 (0.0) [0.0 to 41.0]

5. Primary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with AEs leading to discontinuation of study intervention was reported for each arm.
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 8 | 10 | 7
Percentage of participants | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 41.0] | 0.0 (0.0) [0.0 to 36.9] | 0.0 (0.0) [0.0 to 30.8] | 0.0 (0.0) [0.0 to 41.0]

6. Secondary Outcome: Plasma Concentrations of Ceftolozane
Description: The plasma concentrations of ceftolozane were determined in each group. Blood samples were collected at pre-specified timepoints to determine the plasma concentrations of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: The analysis population consisted of participants who received at least 1 dose of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of ceftolozane.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 6 | 7 | 10 | 7
mg/L
  1 hr post start of infusion | 93.0 (18.9) [lower limit 18.9] | 70.3 (28.6) [lower limit 28.6] | 67.6 (46.9) [lower limit 46.9] | 54.3 (203) [lower limit 203] | 78.5 (19.0) [lower limit 19.0]
  4-5 hrs post start of infusion | 18.8 (20.1) [lower limit 20.1] | 13.4 (55.6) [lower limit 55.6] | 10.5 (52.4) [lower limit 52.4] | 17.6 (83.2) [lower limit 83.2] | 31.8 (45.8) [lower limit 45.8]
  7-8 hrs post start of infusion | 6.61 (27.2) [lower limit 27.2] | 4.53 (53.1) [lower limit 53.1] | 2.79 (59.9) [lower limit 59.9] | 6.84 (172) [lower limit 172] | 19.2 (48.9) [lower limit 48.9]

7. Secondary Outcome: Area Under the Concentration-time Curve of an 8-hour Dosing Interval (AUC0-8) of Plasma Ceftolozane
Description: AUC0-8 was defined as a measure of ceftolozane exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected at pre-specified timepoints to determine the AUC0-8 of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: The analysis population consisted of participants who received at least 6 doses of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of ceftolozane.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
μg*hr/mL | 260 (18.4) [lower limit 18.4] | 230 (27.2) [lower limit 27.2] | 202 (22.5) [lower limit 22.5] | 282 (42.8) [lower limit 42.8] | 360 (29.7) [lower limit 29.7]

8. Secondary Outcome: Maximum Observed Concentration During a Dosage Interval (Cmax) of Plasma Ceftolozane
Description: Cmax was defined as the maximum concentration of ceftolozane observed in plasma. Blood samples were collected at pre-specified timepoints to determine the Cmax of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
μg/mL | 116 (17.8) [lower limit 17.8] | 121 (22.7) [lower limit 22.7] | 107 (15.9) [lower limit 15.9] | 113 (18.9) [lower limit 18.9] | 107 (16.0) [lower limit 16.0]

9. Secondary Outcome: Elimination Half-life (t1/2) of Plasma Ceftolozane
Description: Elimination half-life (t1/2) was defined as the time needed to reduce the level of ceftolozane in the blood by one-half (1/2). Blood samples collected at pre-specified timepoints were used to determine the apparent terminal half-life (t1/2) of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
Hours | 1.87 (8.60) [lower limit 8.60] | 1.56 (16.2) [lower limit 16.2] | 1.33 (15.7) [lower limit 15.7] | 1.79 (39.2) [lower limit 39.2] | 2.60 (24.6) [lower limit 24.6]

10. Secondary Outcome: Clearance (CL) of Plasma Ceftolozane
Description: CL was defined as the total clearance of ceftolozane in plasma over time, assessed as the rate at which ceftolozane was removed from the plasma. Blood samples were collected at pre-specified timepoints to determine the CL of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
L/hr | 7.68 (18.4) [lower limit 18.4] | 4.95 (53.3) [lower limit 53.3] | 2.54 (36.1) [lower limit 36.1] | 0.919 (62.1) [lower limit 62.1] | 0.378 (57.5) [lower limit 57.5]

11. Secondary Outcome: Volume of Distribution (Vd) of Plasma Ceftolozane
Description: Vd was defined as the distributed volume of study drug in plasma at steady state. It is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of the drug. Blood samples were collected at pre-specified timepoints to determine the Vd of ceftolozane in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: The analysis population consisted of participants who received at least 6 doses of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of ceftolozane or tazobactam.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
Liters | 16.2 (18.8) [lower limit 18.8] | 8.35 (50.0) [lower limit 50.0] | 3.97 (17.0) [lower limit 17.0] | 2.13 (36.3) [lower limit 36.3] | 1.36 (34.8) [lower limit 34.8]

12. Secondary Outcome: Plasma Concentrations of Tazobactam
Description: The plasma concentrations of tazobactam were determined in each group. Blood samples were collected at pre-specified timepoints to determine the plasma concentrations of tazobactam in participants receiving ceftolozane/tazobactam. No data were calculated for a timepoint if >50% of samples were below limit of quantification (BLOQ).
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: The analysis population consisted of participants who received at least 1 dose of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of tazobactam.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 6 | 7 | 10 | 7
mg/L
  1 hr post start of infusion | 18.6 (22.4) | 15.5 (43.0) | 15.0 (66.6) | 10.2 (747) | 22.2 (35.5)
  4-5 hrs post start of infusion | 0.876 (38.3) | 0.788 (157) | 0.404 (122) | 0.844 (349) | 3.38 (88.6)
  7-8 hrs post start of infusion | 0.152 (68.4) | 0.181 (183) | NA (NA) — NA= Plasma concentration was not calculated because >50% of samples were BLOQ. | 0.261 (372) | 0.895 (122)

13. Secondary Outcome: Area Under the Concentration-time Curve of an 8-hour Dosing Interval (AUC0-8) of Plasma Tazobactam
Description: AUC0-8 was defined as a measure of tazobactam exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected at pre-specified timepoints to determine the AUC0-8 of tazobactam in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: The analysis population consisted of participants who received at least 6 doses of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of tazobactam.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
μg*hr/mL | 46.7 (25.5) [lower limit 25.5] | 50.1 (42.7) [lower limit 42.7] | 42.7 (33.8) [lower limit 33.8] | 58.3 (50.5) [lower limit 50.5] | 72.5 (35.0) [lower limit 35.0]

14. Secondary Outcome: Maximum Observed Concentration During a Dosage Interval (Cmax) of Plasma Tazobactam
Description: Cmax was defined as the maximum concentration of tazobactam observed in plasma. Blood samples were collected at pre-specified timepoints to determine the Cmax of tazobactam in participants receiving ceftolozane/tazobactam. The analysis population consisted of participants who received at least 6 doses of ceftolozane/tazobactam and had at least 1 quantifiable plasma concentration of tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
μg/mL | 36.7 (29.6) [lower limit 29.6] | 39.4 (34.1) [lower limit 34.1] | 34.2 (24.5) [lower limit 24.5] | 38.1 (29.1) [lower limit 29.1] | 37.9 (14.5) [lower limit 14.5]

15. Secondary Outcome: Elimination Half-life (t1/2) of Plasma Tazobactam
Description: Elimination half-life (t1/2) was defined as the time needed to reduce the level of tazobactam in the blood by one-half (1/2). Blood samples collected at pre-specified timepoints were used to determine the apparent terminal half-life (t1/2) of tazobactam in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
Hours | 1.07 (6.59) [lower limit 6.59] | 0.932 (27.8) [lower limit 27.8] | 0.748 (22.9) [lower limit 22.9] | 0.930 (38.9) [lower limit 38.9] | 1.23 (31.6) [lower limit 31.6]

16. Secondary Outcome: Clearance (CL) of Plasma Tazobactam
Description: CL was defined as the total clearance of tazobactam in plasma over time, assessed as the rate at which tazobactam was removed from the plasma. Blood samples were collected at pre-specified timepoints to determine the CL of tazobactam in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
L/hr | 21.4 (25.5) [lower limit 25.5] | 11.4 (67.6) [lower limit 67.6] | 6.00 (45.9) [lower limit 45.9] | 2.22 (68.5) [lower limit 68.5] | 0.938 (58.2) [lower limit 58.2]

17. Secondary Outcome: Volume of Distribution (Vd) of Plasma Tazobactam
Description: Vd is defined as the distributed volume of study drug in plasma at steady state. It is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of the drug. Blood samples were collected at pre-specified timepoints to determine the Vd of tazobactam in participants receiving ceftolozane/tazobactam.
Time Frame: Day 3: 1, between 4-5, and between 7-8 hours post start of infusion
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Group 1: Ceftolozane/Tazobactam 12 to <18 Years of Age | Group 2: Ceftolozane/Tazobactam 7 to <12 Years of Age | Group 3: Ceftolozane/Tazobactam 2 to <7 Years of Age | Group 4: Ceftolozane/Tazobactam 3 Months to <2 Years of Age | Group 5: Ceftolozane/Tazobactam Birth to <3 Months of Age
Number analyzed (Participants) | 8 | 7 | 7 | 10 | 7
Liters | 15.2 (37.9) [lower limit 37.9] | 7.71 (74.6) [lower limit 74.6] | 3.34 (17.3) [lower limit 17.3] | 2.07 (32.5) [lower limit 32.5] | 1.38 (23.7) [lower limit 23.7]

ADVERSE EVENTS:
Time Frame: Up to approximately 31 days
Description: Analysis population for All-cause mortality consists of all enrolled participants. Serious and Other adverse events include all participants who received any dose (including partial doses) of ceftolozane/tazobactam.
Groups:
- Group 1: 12 to <18 Years: Participants 12 to <18 years of age with nosocomial pneumonia received intravenous (IV) ceftolozane 2g and tazobactam 1g every 8 hours for 8-14 days.
- Group 2: 7 to <12 Years: Participants 7 to <12 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 3: 2 to <7 Years: Participants 2 to <7 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 4: 3 Months to <2 Years: Participants 3 months to <2 years of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and tazobactam 20 mg/kg every 8 hours for 8-14 days.
- Group 5: Birth to <3 Months: Participants from birth to <3 months of age with nosocomial pneumonia received IV ceftolozane 40 mg/kg and 20 mg/kg tazobactam every 8 hours for 8-14 days.
Arm/Group | Group 1: 12 to <18 Years | Group 2: 7 to <12 Years | Group 3: 2 to <7 Years | Group 4: 3 Months to <2 Years | Group 5: Birth to <3 Months
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8 | 2/10 | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/7 | 0/8 | 3/10 | 2/7
Other Adverse Events (participants affected / at risk) | 4/8 | 5/7 | 6/8 | 9/10 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 12 to <18 Years (N=8) | Group 2: 7 to <12 Years (N=7) | Group 3: 2 to <7 Years (N=8) | Group 4: 3 Months to <2 Years (N=10) | Group 5: Birth to <3 Months (N=7)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial depression (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Omentitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 12 to <18 Years (N=8) | Group 2: 7 to <12 Years (N=7) | Group 3: 2 to <7 Years (N=8) | Group 4: 3 Months to <2 Years (N=10) | Group 5: Birth to <3 Months (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2)
Withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Base excess decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04223752/Prot_SAP_000.pdf